CLINICAL TRIAL: NCT01050322
Title: A Randomized Open-Label, Phase II Study of Lapatinib-capecitabine or Lapatinib-vinorelbine or Lapatinib/Gemcitabine in Subjects With Her2/Neu Amplified Metastatic Breast Cancer Patients Progression After Taxanes Treatment
Brief Title: Safety Study in Subjects With Metastatic Breast Cancer Who Progressed After Taxanes Treatment.
Acronym: GLICO-0801
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLICO-0801
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2010-11

CONDITIONS: BRMS1; Performance Status Zero to Two for Beginning the Study; Patient With a Maximum of One Chemotherapy; Patient With Progression After Taxanes
Keywords: receptor HER two positive; lapatinib; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Capecitabine Lapatinib (Active Comparator): The starting dose of capecitabine is 2000 mg/m2/day, to be divided and given twice daily orally, 12 hours apart, for 14 days, every 21 days. A daily dose of Lapatinib is 5 tablets (1250 mg of Lapatinib) taken approximately at the same time each day.
  Interventions: Drug: Lapatinib Capecitabine
- Vinorelbine Lapatinib (Experimental): The starting dose of vinorelbine is 25 mg/m2/ IV days 1 and 8, every 21 days. A daily dose of Lapatinib is 5 tablets (1250 mg of Lapatinib) taken approximately at the same time each day.
  Interventions: Drug: Lapatinib Vinorelbine
- Gemcitabine Lapatinib (Experimental): The starting dose of gemcitabine is 1000mg/m2/ IV days 1 and 8, every 21 days. A daily dose of Lapatinib is 5 tablets (1250 mg of Lapatinib) taken approximately at the same time each day.
  Interventions: Drug: Gemcitabine Lapatinib

INTERVENTIONS:
Drug: Lapatinib Vinorelbine — The starting dose of vinorelbine is 25 mg/m2/ IV days 1 and 8, every 21 days. A daily dose of Lapatinib is 5 tablets (1250 mg of Lapatinib) taken approximately at the same time each day.
  Arms: Vinorelbine Lapatinib
Drug: Lapatinib Capecitabine — The starting dose of capecitabine is 2000 mg/m2/day, to be divided and given twice daily orally, 12 hours apart, for 14 days, every 21 days. A daily dose of Lapatinib is 5 tablets (1250 mg of Lapatinib) taken approximately at the same time each day.
  Arms: Capecitabine Lapatinib
Drug: Gemcitabine Lapatinib — The starting dose of gemcitabine is 1000mg/m2/ IV days 1 and 8, every 21 days. A daily dose of Lapatinib is 5 tablets (1250 mg of Lapatinib) taken approximately at the same time each day.
  Arms: Gemcitabine Lapatinib

SUMMARY:
Despite these initial positive signals in recent statistics, breast cancer continues to claim a substantial number of lives approximately 500,000 deaths worldwide in 2005 Thus the current treatment paradigm - surgery, radiation and systemic chemo and or hormonal therapy and biological therapies -still fails to cure a significant number of women with early breast cancer and new treatment strategies are needed to improve current results both in early and advance disease.

Recurrent or metastatic breast cancer is an incurable malignancy with a median survival of 20-24 months [Hortobagyi , 1998] and this has not changed significantly over the last decade with fewer than 20% of patients still alive at 5 years after a diagnosis of recurrence. Although there have been small improvements in survival with the new therapies, metastatic breast cancer remains an incurable and, ultimately, fatal disease. The introduction of novel combination therapies have the potential to target different pathways in the cancer cell, leading to improved efficacy. Further studies to optimize combination therapy, while ameliorating AEs, are critically important to patients with metastatic breast cancer.

Lapatinib is an oral tyrosine kinase inhibitor which potently inhibits both EGFR and HER2[Spector, 2005]. Lapatinib in combination with capecitabine is approved in more than 20 countries for the treatment of patients with advanced or metastatic breast cancer whose tumors overexpress HER2. All patients in the study leading to the lapatinib approval had received prior therapy including an anthracycline, a taxane, and trastuzumab.

The relevance of the HER2/neu target in breast cancer, combined with the promising preclinical and clinical data regarding the use of lapatinib, provide the rationale for a formal evaluation of this agent combined with other non taxane agents as gemcitabine or vinorelbine after progression on taxanes and trastuzumab based therapies in metastatic disease setting as these chemotherapy options are used in daily practice in this subset of patients.

This is a randomized phase II, open label,multicentric , international, 3 arms treatment study in patients with confirmed HER2+ metastatic breast cancer after taxane progression . The main objective is to investigate the (CBR) and safety in 3 different combinations of Lapatinib therapy (plus capecitabine or gemcitabine or vinorelbine) and to determine whether either, or both, of Lapatinib /Vinorelbine or Lapatinib/Gemcitabine can be considered a reasonable alternative to the established Lapatinib/Capecitabine standard combination . The decision as to whether to study either of the new combinations further will be based on both the toxicity and the efficacy profiles.

DETAILED DESCRIPTION:
In areas where trastuzumab is available with no barriers to access, all patients must have received trastuzumab in the adjuvant or metastatic setting . However, in countries where trastuzumab is not approved or is not available to patients due to reimbursement or other considerations, trastuzumab naïve patients are allowed considering the efficacy data of Lapatinib in this subset of patients.

This trial uses a design to ensure a selection of one or more of the better treatment combination for additional clinical Approximately (165), who meet the criteria for efficacy analysis as defined, will be enrolled in the study in a single stage process. The sample size will be accrued in 16 months, with further follow-up for a 24 months study period from randomization or until progression.

The study includes a Screening/Baseline Period, a Treatment Period and a post-treatment Follow-Up Period. Patients will continue to receive investigational products until disease progression or early discontinuation from investigational product for other reasons. Patients who discontinue investigational product(s) without disease progression will continue to be evaluated for efficacy until progression or until receiving the first subsequent anti-cancer therapy. Once progression is documented, all patients will be followed for survival at approximately 3-month intervals until death.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained according to local ethical committee requirements.
2. Subjects must be older than 18 years old.
3. Histologically confirmed invasive adenocarcinoma of the breast which is stage IIIb, stage IIIc with T4 lesion, or stage IV disease [according to AJCC 6th edition]
4. Documented progression after taxane based treatment for ErbB2 positive patients for 1st line metastatic breast cancer or documented progression after taxane based regimens as adjuvant or neo-adjuvant therapy. Patients may have had a maximum of one prior treatment with a chemotherapy regimen for metastatic disease.
5. Patients must have at least 1 measurable lesion defined by RECIST as follows:

   * X-ray, physical exam > 20 mm.
   * Conventional CT scan > 20 mm.
   * Spiral CT scan > 10 mm.
   * Measurable lesions must be outside a previous radiotherapy field if they are the sole site of disease.
6. Local laboratory confirmed HER2/neu over expressing and/or amplified disease in the invasive component of the primary or metastatic lesion as defined by at least one of the following based local results:

   * 3+ overexpression by IHC (> 30% of invasive tumour cells).
   * 2+ or 3+ (in 30% or < % of neoplastic cells) over expression by IHC AND in situ hybridization (FISH/CISH) test demonstrating HER2 gene amplification.
   * HER2 gene amplification by FISH or CISH. (> 6 HER2 gene copies per nucleus, or a FISH ratio (HER2 gene copies to chromosome 17 signals) of > than 2.2.
7. Prior therapy must have included a taxane regimen. Patients must have received either:

   * Prior adjuvant treatments with taxanes-containing chemotherapy regimens providing that at least 6 months has elapsed from the last dose of adjuvant or neoadjuvant chemotherapy and all treatment related adverse events are < grade 1 at the time of randomization; OR
   * Prior treatment with taxane based chemotherapeutic regimens for first line metastatic breast cancer or prior taxane based neoadjuvant regimens for locally advanced disease providing that at least 4 weeks has elapsed since the last dose of therapy for metastatic disease and all treatment related adverse events are < grade 1 at the time of randomization.
8. In regions where trastuzumab is available with no barriers to access, patients must have also received prior trastuzumab alone or in combination with chemotherapy in order to be eligible as follows:

   * Prior treatment with Trastuzumab includes only first line metastatic setting; OR
   * Prior trastuzumab treatment in neoadjuvant / adjuvant setting provided that at least 6 months has elapsed from last dose of adjuvant / neoadjuvant Trastuzumab , and all treatment related adverse events are < grade 1 at the time of randomization.
9. Prior treatment with anthracyclines in the adjuvant or first line metastatic setting are permitted provided that therapy has been discontinued before randomization, and all treatment related adverse events are < grade 1 at the time of randomization.
10. Prior treatment with endocrine therapy in the adjuvant or metastatic setting are permitted provided that therapy has been discontinued before randomization, and all treatment related adverse events are < grade 1 at the time of randomization.
11. Prior treatments with radiation therapy for palliative management of metastatic disease , to a limited area (e.g., palliative treatment for painful disease) other than the sole site of measurable and assessable disease is allowed however, subjects must have completed treatment at least 4 weeks of the last dose of radiotherapy prior to starting study drugs, and must have recovered from all treatment-related toxicities prior to Day 1.

11. Life expectancy of at least 6 months.

12. ECOG PS 0-2.

13. Patients must have normal organ and marrow function measured within 14 days prior to randomization as defined below:

* System Laboratory Values
* Hematologic
* Absolute neutrophil count (ANC) > 1.5 X 109/L
* Hemoglobin1 > 9 g/dL
* Platelets > 100 X 109/L
* Hepatic
* Albumin > 2.5 gr /dl
* Total bilirubin > 1.5 X upper limit of normal (ULN)
* AST and ALT > 2.5 X ULN
* Renal
* Serum Creatinine > 1.5 mg/dL o 132.6 micromol/L
* Or, if serum creatinine > 1.5 mg/dL, Calculated creatinine clearance > 50 mL/min
* Patients may not have had a transfusion within 7 days of screening assessment

  14. CT head/MRI within 4 weeks prior to randomization.

  15. Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to registration.

  16. Patients must have at least 1 measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST, Therasse, 2000). Measurable lesions may be in the field of prior adjuvant irradiation. However, there must be at least a 4 week period between the last radiation treatment and the baseline scan documenting disease status. Documented progression of the irradiated lesion is also required for the lesion to be considered measurable.

  17. Subjects must have a cardiac ejection fraction within the institutional range of normal as measured by ECHO (echocardiogram) or alternatively by MUGA (Multigated Acquisition) scan. Cardiac ejection fraction > 50% and within the institutional range of normal as demonstrated by echocardiogram or alternatively by MUGA scan within 4 weeks of randomization Subjects with known uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure are NOT eligible;

  18. Subjects must complete all screening assessments as outlined in the protocol.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Prior therapy with other anti Erbb1 or antiErbB2 targeted agent rather than Trastuzumab only limited to 1st line treatment of metastatic disease OR as adjuvant/neoadjuvant therapy.
3. Prior exposure to gemcitabine , vinorelbine and capecitabine for 1st line treatment of recurrent-metastatic disease OR as adjuvant / neoadjuvant therapy.
4. Treatment in the 14 days prior to randomization with anti-cancer therapy (tumor embolization, chemotherapy , immunotherapy, biological therapy, or hormonal therapy) or treatment with mitomycin within 6 weeks prior to randomization. Such treatment may not be resumed or begun after study entry. Note: Patients receiving bisphosphonate therapy prior to randomization may continue for the duration of study participation, however bisphosphonates should not be initiated following study entry.

   Prophylactic use of bisphosphonates in subjects without bone disease is not permitted, except for the treatment of osteoporosis.
5. Active CNS metastases.
6. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, serious non-healing wound/ulcer/bone fracture, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
8. Have current active hepatic or biliary disease(with exception of patients with Gilbert syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
9. History of other malignancy. Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
10. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
11. Concurrent treatment with an investigational agent or participation in another clinical trial.
12. Used an investigational drug within 30 days or 3 half-lives, whichever is longer, preceding the first dose of therapy.
13. History of immediate or delayed hypersensitivity or idiosyncrasy to drugs chemically parented to Lapatinib or navelbine or capecitabine or gemcitabine and its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate | 6 months

SECONDARY OUTCOMES:
Evaluate: PFS and OS each treatment arm. Determine ORR and duration of response of each treatment. Incidence AE,SAEs Determine quale and quantic toxicities associated with LAPATINIB when administered with other chemotherapy different capecitabine. | 6 months

CONTACTS AND LOCATIONS:
Locations (18):
- Argentina (8):
  - Dr. Guillermo Lerzo, Buenos Aires
  - Dr. Eduardo Richardet, Córdoba
  - Dr. Adolfo Capó, Mendoza
  - Dr. Juan Lacava, Neuquén
  - Dra. Mirta Varela, Quilmes
  - Dr. Luis Fein, Rosario
  - Dr. Jose Zarba, San Miguel de Tucumán
  - Dr. Cesar Blajman, Santa Fe
- Brazil (9):
  - Dr. Carlos Alberto Sampaio, Salvador, Estado de Bahia
  - Dr. José Bines, Rio de Janeiro, Rio de Janeiro
  - Dr. Carlos Barrios, Porto Alegre, Rio Grande do Sul
  - Dra. Yeni Veronica Neron, Florianópolis, Santa Catarina
  - Dr. Gustavo Ismael, Jaú, São Paulo
  - Dra. Patricia Xavier Santi, Santo André, São Paulo
  - Dr. Max Mano, São Paulo, São Paulo
  - Dr. Marcello Fanelli, São Paulo, São Paulo
  - Dra. Célia Tosselo de Oliveira, São Paulo, São Paulo
- Dra. Silvia Neciosup, Lima, Peru, Peru

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241